CLINICAL TRIAL: NCT03427255
Title: A Cognitive Behavioral Group Program-plus for Women With Dyspareunia: A Randomized Waiting List Controlled Multi-center Trial of Efficacy
Brief Title: CBT Group Treatment for Women With Dyspareunia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Örebro University, Sweden (Other)
Collaborators: Leiden University Medical Center (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBT group program-plus
Record Dates: First submitted 2017-12-01; First posted 2018-02-09 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Dyspareunia
Keywords: superficial dyspareunia; CBT
MeSH Terms: conditions — Dyspareunia; Color Vision Defects

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with a waiting list condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT group treatment (Active Comparator): CBT group treatment-plus involving partners: 10 group sessions and 3 couple sessions
  Interventions: Behavioral: CBT group treatment-plus
- Waiting list (Other): Six months waiting-list control condition.
  Interventions: Behavioral: CBT group treatment-plus; Other: Waiting-list control condition

INTERVENTIONS:
Behavioral: CBT group treatment-plus — The CBT group program-plus consists of 3 1- hr CBT couple sessions and 10 2-hr CBT group sessions over a period of 6 months. The manualized treatment comprise, pain- and sexual education, relaxation and gradual exposure exercises as well as sensate focus and sexual communication exercises for the couple. 6-8 women participate in each group. Two psychologists conduct the couple and group sessions.
Other: Waiting-list control condition — Waiting-list control condition during length of active treatment (6 months).
  Arms: Waiting list

SUMMARY:
The current study will employ a group CBT treatment program of 10 group sessions and 3 individual couple sessions targeting the thoughts, emotions, behaviors and couple interactions associated with the experience of dyspareunia. Women with superficial dyspareunia and their partners will be randomized to the CBT group program-plus or a waiting list control period at one treatment location in Sweden and two treatment locations in the Netherlands. The waiting-list control period will be comparable to the treatment duration of six months.

It is hypothesized that the group program-plus is more effective in improving pain during intercourse in women with superficial dyspareunia compared to women on a waiting-list control period.

DETAILED DESCRIPTION:
Rationale:

Superficial dyspareunia, a frequent form of chronic genital pain, is associated with decreased sexual function for afflicted women, as well as impoverished sexual satisfaction for women and their partners. While recent research has showed that cognitive-behavioral therapy (CBT) interventions have effects in regards to reducing pain, enhancing sexual function and improving relational aspects, randomized controlled trials are still sparse. Despite recommendations in the literature to include the partner in the CBT treatment targeted at improving pain and sexuality outcomes, there are no published randomized CBT controlled trials incorporating the partner in the treatment.

Primary objective: To evaluate whether the group program-plus improves pain during intercourse in women with superficial dyspareunia compared to women in a waiting-list control condition.

Secondary Objective(s): are to evaluate a) women (and partners) sexuality (sexual function, distress & satisfaction), b) women's psychological adjustment (negative and positive penetration beliefs, pain/penetration coping behavior); c) relationship factors (partner responses and relationship satisfaction), and whether an improvement in pain during intercourse is moderated by pre-treatment patient characteristics, such as age, sexual functioning, relationship satisfaction, abuse history, and mediated by a) reduction of negative penetration beliefs, avoidance behavior and/or improvement in positive penetration beliefs and sexual function (i.e. sexual arousal).

Study design:

Eligible women and their partners in one of the participating centers (n=3, in two countries) will be randomized to either the CBT group program-plus or waiting-list control group (WLC), using a block randomization design stratified for each center. The waiting-list period of 6 months is comparable to the period from the start of the active treatment until the post-treatment measurement. After the WLC, the patients from the WLC will receive the active treatment. Data of these participants will be included in the repeated measures analyses to test the temporal stability of treatment gains. Within-subjects repeated measures comparisons will be conducted for data of participants and their partners at pre-treatment, post-treatment, follow-up at 3 months and 6 months following treatment termination. In addition, participants complete monthly questionnaires at home during the first 6 months. Participants in the active treatment group will also complete weekly measures. These extra measurement are necessary for the mediation analyses. The total study duration (including follow-up) for the participants and their partners is 12-18 months.

Intervention:

The CBT group program-plus consists of 3 1-hr CBT couple sessions and 10 2-hr CBT group sessions over a period of 6 months. The manualized treatment comprise, pain- and sexual education, relaxation and gradual exposure exercises as well as sensate focus and sexual communication exercises for the couple. 6-8 women participate in each group. Two psychologists will conduct the couple and group sessions.

ELIGIBILITY:
Inclusion Criteria:

* woman
* 18-45 years old
* in a heterosexual relationship for at least 3 months
* diagnosis of superficial dyspareunia (in accordance to DSM5) with no apparent ongoing physical cause to the condition (i.e. ongoing infections).
* past experience of a successful intercourse
* attempted intercourse during the last year

Exclusion Criteria:

* reporting to never have had full intercourse at any time in life
* partner not willing to participate in the study
* major affective disorder, psychotic disorder, substance-related disorder or post traumatic-stress disorder related to the genitals (e.g., as a sequel to sexual abuse) according to DSM-5 criteria
* being pregnant
* gone through child delivery during the last year
* not speaking Dutch or Swedish well enough to participate in assessment and treatment
* receiving concurrent psychological therapy or physiotherapy for superficial dyspareunia during CBT or WLC period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean level of pain during penile/vaginal intercourse (PI) | 6 months; 9 months; 12 months
  Pain intensity is measured on a scale between 0-10

SECONDARY OUTCOMES:
Penetration behavior questionnaire (PBQ) | 6 months; 9 months; 12 months
  The PBQ has seven questions inquiring about the woman's experience during the last month with the following aspects of vaginal penetration: full vaginal penetration with the penis of the partner, self-insertion in the vagina of one finger by the woman, self-insertion in the vagina of two fingers by the woman, insertion in the vagina of one finger by the partner, insertion in the vagina of two fingers by the partner, and self-insertion in the vagina of another object (such as a tampon or a dildo) by the woman and by the partner. Answering categories are as follows: (a) not attempted; (b) attempted, but unsuccessful; (c) attempted and sometimes successful; and (d) attempted and always successful. The total of the scale is calculated and ranges between 4-28.
Genital pain rating questionnaire (GPQ) | 6 months; 9 months; 12 months
  Genital pain experienced by touch and penetration of the vagina will be assessed with the 7- item Genital Pain rating Questionnaire (GPQ). Response categories vary from 0 (not at all) to 10 (worst pain imaginable). The questionnaire consist of two sub-scales: the first sub-scale 'pain on touch and finger insertion'' consists of 6 items (pain by touch of the vulva by the patient herself, pain by touch of the vulva by the patient's partner, pain during insertion of one/two own finger(s) into the vagina, and pain during insertion of one/two finger(s) of the patient's partner) into the vagina. The range of the sub-scale is 0-60. The second sub-scale is 1 item related to pain during intercourse (0-10).
Female Sexual Function Index (FSFI) | 6 months; 9 months; 12 months
  Female Sexual functioning will be assessed with the 19-item Female Sexual Function Index (FSFI). It covers six domains of sexual functioning: sexual desire, sexual arousal, lubrication, orgasm, sexual satisfaction, and sexual pain. The answers are given on a Likert scale ranging from 0 or 1 to 5, depending on item. For the current study, the total FSFI score will be used, excluding the three items on sexual pain, which gives an indication of the sexual functioning during the past four weeks. The total score ranges between 2-30 with higher scores indicating higher sexual function.
Female Sexual Distress scale (FSDS) | 6 months; 9 months; 12 months
  Sexual related personal distress will be assessed with the 12-item Female Sexual Distress scale (FSDS). Questions are answered on a 0-4 Likert scale and the total score ranges from 0-48 with higher scores indicating higher sexual distress.
Global Measure of Sexual Satisfaction Scale (GMSEX) | 6 months; 9 months; 12 months
  Sexual satisfaction will be assessed with the 5-item Global Measure of Sexual Satisfaction Scale (GMSEX). GMSEX consist of five 7-point dimensions of sexual satisfaction ranging from "Good" to "Bad", "Pleasant" to "Unpleasant", "Positive" to "Negative", "Satisfying" to "Unsatisfying", and "Valuable" to "Worthless". Total scores range from 5-35, with higher scores indicating greater sexual satisfaction.
Vaginal Penetration Cognition Questionnaire (VPCQ) | 6 months; 9 months; 12 months
  Positive and negative cognitions and beliefs regarding vaginal penetration will be assessed with the 22-item Vaginal Penetration Cognition Questionnaire (VPCQ). The VPCQ is a 22-item self-report measure using positive and negative statements about vaginal penetration and is answered on a 7-point Likert scale. Possible answers range from "0 = not at all applicable" to "6 = very strongly applicable." The VPCQ consists of 5 subscales: Control Beliefs (4 items), Catastrophic and Pain Beliefs (5 items), Self-Image Beliefs (6 items), Positive Beliefs (5 items), and Genital Incompatibility Beliefs (2 items).
Painful Intercourse Self-Efficacy Scale (PISES) | 6 months; 9 months; 12 months
  Pain self-efficacy beliefs will be assessed using the 20-item Painful Intercourse Self-Efficacy Scale (PISES), it consists of three sub-scales: self-efficacy for controlling pain during intercourse, for sexual function, and for other symptoms. Answers are given on a 10-point scale ranging from (10) very uncertain to (100) very certain.
CHAMP Sexual Pain Coping Scale (CSPCS) | 6 months; 9 months; 12 months
  Avoidance and endurance coping behaviors during penetration will be assessed with the 12-item CHAMP Sexual Pain Coping Scale (CSPCS). This measure consists of three sub-scales: avoidance, endurance and alternative strategies. Respondents rate their agreement of each statement between 1 ("Never true") and 7 ("Always true"). Total scores range from 4-28 on each sub-scale.
Maudsley Marital Questionnaire (MMQ) | 6 months; 9 months; 12 months
  Relationship satisfaction will be assessed with the 10 items of the marital dissatisfaction subscale of the Maudsley Marital Questionnaire MMQ. Possible range 0-80 with higher scores indicating greater dissatisfaction.
Approach and Avoidance Sexual Goals (AASG) | 6 months; 9 months; 12 months
  To assess sexual motives and goals the 15-item Approach and Avoidance Sexual Goals (AASG) measure will be used. Participants can rate the importance of 9 approach and 6 interpersonal goals in influencing their decision to engage in sex on a 7 point scale.

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 6 months; 9 months; 12 months
  Symptoms of depression will be assessed with the 9 item Patient Health Questionnaire (PHQ-9). The answers are given on a scale between 0-3 and total scores ranges between 0-27 with higher scores indicative of higher symptoms of depression.
Generalized Anxiety Disorder-7 (GAD-7) | 6 months; 9 months; 12 months
  Symptoms of anxiety will be assessed with the 7 item generalized anxiety disorder-7 (GAD-7). The answers are given on a scale between 0-3 and total scores ranges between 0-21 with higher scores indicative of higher symptoms of anxiety.
International Index of Erectile Dysfunction (IIEF) | 6 months; 9 months; 12 months
  Male sexual function will be assessed with the 15 items of the International Index of Erectile Function (IIEF) which is a widely used, multi-dimensional self-report instrument for the evaluation of male sexual function. The answers are given on a Likert scale ranging from 0 or 1 to 5, depending on item. For the current study, the total IIEF score will be used, which gives an indication of the sexual functioning during the past four weeks. The total score ranges between 2-30 with higher scores indicating higher sexual function.
Male Sexual Distress Scale (MSDS) | 6 months; 9 months; 12 months
  Sexual related personal distress will be assessed with the 12-item Female Sexual Distress scale (FSDS). Because the FSDS does not contain gender specific items, the measure has also successfully been administered to male participants. Questions are answered on a 0-4 Likert scale and the total score ranges from 0-48 with higher scores indicating higher sexual distress.
Perceived treatment improvement and satisfaction | 6 months; 9 months; 12 months
  Self-reported improvement (scale of 0 (worse) to 5 (complete cure)) and treatment satisfaction (scale of 0 (completely dissatisfied) to 10 (completely satisfied)) are measured to assess the clinical significance of results.
EuroQual5 (EQ-5D) | 6 months; 9 months; 12 months
  Is used to assess general function. The visual analogue scale (VAS) of the EQ-5D will be used as a quantitative measure of health as judged by the woman and her partner ranging between 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Ida K Flink, PhD, Principal Investigator — Örebro University, Sweden; Moniek M ter Kuile, PhD, Principal Investigator — Leiden University Medical Center
Locations (3):
- Netherlands (2):
  - Leiden University Medical Center, Department of Gynecology, Leiden
  - Maastricht Universiy Medical Center (MUMC), Maastricht
- Center for Health and Medical Psychology (CHAMP) Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No